CLINICAL TRIAL: NCT01772147
Title: A Multicenter, Randomized, Double-blind, Parallelgroup Study to Evaluate the Efficacy and Safety of the Addition of Umeclidinium Bromide Inhalation Powder (62.5mcg) Once-daily to Fluticasone Propionate/Salmeterol (250/50mcg) Twice-daily, Umeclidinium Bromide Inhalation Powder (125mcg) Once-daily to Fluticasone Propionate/Salmeterol (250/50mcg) Twice-daily Versus Placebo to Fluticasone Propionate/Salmeterol (250/50mcg) Twice-daily Over 12 Weeks in Subjects With COPD.
Brief Title: Efficacy and Safety of the Addition of Fluticasone Propionate/Salmeterol (250/50mcg) Twice-daily to 2 Doses of Umeclidinium Bromide Inhalation Powder (62.5 or 125mcg) Once-daily Over 12 Weeks.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116136
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umeclidinium bromide (Experimental): Long-acting muscarinic antagonist (LAMA)
  Interventions: Drug: Umeclidinium bromide 62.5mcg; Drug: Umeclidinium bromide 125mcg
- Fluticasone propionate/Salmeterol (Active Comparator): Inhaled corticosteroid (ICS)/Long-acting beta agonist (LABA)
  Interventions: Drug: Fluticasone propionate 250mcg/Salmeterol 50mcg

INTERVENTIONS:
Drug: Umeclidinium bromide 62.5mcg — Inhalation powder
  Arms: Umeclidinium bromide
Drug: Umeclidinium bromide 125mcg — Inhalation powder
  Arms: Umeclidinium bromide
Drug: Fluticasone propionate 250mcg/Salmeterol 50mcg — Inhalation powder
  Arms: Fluticasone propionate/Salmeterol

SUMMARY:
The purpose of this 12 week study is to evaluate the effects of the addition of umeclidinium bromide (62.5mcg) once-daily to fluticasone propionate (250/50mcg) twice-daily and umeclidinium bromide (125mcg) once-daily to fluticasone propionate (250/50mcg) twice-daily with placebo when added to fluticasone propionate (250/50mcg) twice-daily on lung function, COPD-related health status assessments and safety in COPD subjects.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group study. Subjects who meet the eligibility criteria at screening and meet the randomization criteria at the end of a 4 week run-in period will enter a 12 week treatment period. There will be a 7 day follow-up period after the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient.
* Informed Consent: A signed and dated written informed consent prior to study participation.
* Age: Subjects 40 years of age or older at Visit 1.
* Gender: Male or female subjects. A female is eligible to enter and participate if of non-child-bearing potential, or if of child bearing potential, has a megative serum pregnancy test at screening, and agrees to one of the acceptable contraceptive methods listed in the protocol, used consistently and correctly.
* Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society.
* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of ≥10 pack-years [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Pipe and/or cigar use cannot be used to calculate pack year history.
* Severity of Disease: A pre and post-albuterol/salbutamol FEV1/FVC ratio of <0.70 and a pre and post-albuterol/salbutamol FEV1 of ≤70% of predicted normal values at Visit 1 (Screening) calculated using Nutrition Health and Examination Survey (NHANES) III reference equations.
* Dyspnea: A score of ≥2 on the mMRC Dyspnea Scale at Visit 1.

Exclusion Criteria:

* -Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: A current diagnosis of asthma.
* Other Respiratory Disorders: Known α-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. A subject who, in the opinion of the investigator, has any other significant respiratory conditions in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease.
* Other Diseases/Abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for <5 years prior to Visit 1 (localized carcinoma of the skin that has been resected for cure is not exclusionary). Significant is defined as any disease that,in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Contraindications: Any history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, sympathomimetic, corticosteroid (intranasal, inhaled or systemic) lactose/milk protein or magnesium stearate, or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the study physician contraindicates study participation or use of an inhaled anticholingeric.
* Hospitalization: Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
* Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Visit 1.
* 12-Lead ECG: An abnormal and significant ECG finding from the 12-lead ECG conducted at Visit 1. Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility. Specific ECG findings that preclude subject eligibility are listed in Appendix 4. The study investigator will determine the medical significance of any ECG abnormalities not listed in Appendix 4.
* Medication Prior to Spirometry: Unable to withhold albuterol/salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
* Medications Prior to Screening: use of certain medications for the protocol-specific times prior to Visit 1.

Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., ≤12 hours per day) is not exclusionary.

* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., albuterol/salbutamol) via nebulized therapy.
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, subinvestigator, study coordinator, or employee of the participating investigator.
* Inability to read: In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a questionnaire.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (42):
- United States (16):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Chile (5):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Concepción, Región Del Biobio
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Talca, Región Metro de Santiago
- Czechia (9):
  - GSK Investigational Site, Karlovy Vary
  - GSK Investigational Site, Kralupy nad Vltavou
  - GSK Investigational Site, Lovosice
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Tábor
  - GSK Investigational Site, Teplice
- Poland (9):
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Grudziądz
  - GSK Investigational Site, Inowrocław
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Ostrów Wielkopolski
  - GSK Investigational Site, Piła
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- South Korea (3):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Seongnam-si, Gyeonggi-do
  - GSK Investigational Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 116136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116136 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 872 participants who met the eligibility criteria at Screening (Visit 1) started a 28-day Run-in Period, in which they received open-label fluticasone propionate and salmeterol (FSC) 250/50 micrograms (µg), prior to being randomized to a 12-week randomized Treatment Period.
Pre-assignment Details: A total of 608 participants were randomized in the study; however, only 606 of these 608 participants were included in the Intent-to-Treat Population, comprised of all participants randomized to treatment who received at least one dose of randomized study medication in the Treatment Period.
Groups:
- Placebo QD + FSC 250/50 µg BID: Participants received placebo once daily (QD) each morning via a dry powder inhaler (DPI) and FSC 250/50 µg twice daily (BID) (one inhalation each morning and one inhalation each evening) via a DPI for 12 weeks.
- UMEC 62.5 µg QD + FSC 250/50 µg BID: Participants received umeclidinium bromide (UMEC) 62.5 µg QD each morning via a DPI and FSC 250/50 µg BID (one inhalation each morning and one inhalation each evening) via a DPI for 12 weeks.
- UMEC 125 µg QD + FSC 250/50 µg BID: Participants received UMEC 125 µg QD each morning via a DPI and FSC 250/50 µg BID (one inhalation each morning and one inhalation each evening) via a DPI for 12 weeks.
Period: Overall Study
Arm/Group | Placebo QD + FSC 250/50 µg BID | UMEC 62.5 µg QD + FSC 250/50 µg BID | UMEC 125 µg QD + FSC 250/50 µg BID
Started | 201 | 203 | 202
Completed | 170 | 178 | 184
Not Completed | 31 | 25 | 18
Not completed — Adverse Event | 13 | 10 | 6
Not completed — Withdrew Consent | 7 | 8 | 4
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Protocol Deviation | 2 | 1 | 1
Not completed — Lack of Efficacy | 8 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Placebo QD + FSC 250/50 µg BID: Participants received placebo QD each morning via a DPI and FSC 250/50 µg BID (one inhalation each morning and one inhalation each evening) via a DPI for 12 weeks.
- UMEC 62.5 µg QD + FSC 250/50 µg BID: Participants received UMEC 62.5 µg QD each morning via a DPI and FSC 250/50 µg BID (one inhalation each morning and one inhalation each evening) via a DPI for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo QD + FSC 250/50 µg BID | UMEC 62.5 µg QD + FSC 250/50 µg BID | UMEC 125 µg QD + FSC 250/50 µg BID | Total
Number analyzed (Participants) | 201 | 203 | 202 | 606
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (7.92) | 64.5 (8.31) | 65.5 (7.89) | 65.2 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 63 | 82 | 223
  Male | 123 | 140 | 120 | 383
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 3 | 5 | 4 | 12
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Japanese/East Asian Heritage/South East Asian | 37 | 33 | 27 | 97
  White | 161 | 164 | 171 | 496

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Trough Forced Expiratory Volume in One Second (FEV1) on Day 85
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Treatment Day 85 is defined as the mean of the FEV1 values obtained 23 and 24 hours after dosing on Treatment Day 84 (i.e., at Week 12). Baseline trough FEV1 is the mean of the two assessments made at -30 and -5 minutes (min) pre-dose on Treatment Day 1. Change from Baseline was calculated as the Day 85 value minus the Baseline value. Analysis was performed using a repeated measures model with covariates of treatment, Baseline (mean of the two assessments made at -30 and -5 min pre-dose on Treatment Day 1), smoking status, day, day by Baseline, and day by treatment interactions.
Time Frame: Baseline and Day 85
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of randomized study medication in the Treatment Period. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo QD + FSC 250/50 µg BID | UMEC 62.5 µg QD + FSC 250/50 µg BID | UMEC 125 µg QD + FSC 250/50 µg BID
Number analyzed (Participants) | 169 | 178 | 183
Liters | -0.001 (0.0136) | 0.126 (0.0133) | 0.147 (0.0132)
Statistical Analysis 1: Comparison: Placebo QD + FSC 250/50 µg BID vs UMEC 62.5 µg QD + FSC 250/50 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.127, 95% CI 2-sided [0.089 to 0.164]
Statistical Analysis 2: Comparison: Placebo QD + FSC 250/50 µg BID vs UMEC 125 µg QD + FSC 250/50 µg BID; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.148, 95% CI 2-sided [0.111 to 0.185]

2. Secondary Outcome: Change From Baseline in Weighted Mean 0-6 Hour FEV1 Obtained Post-dose at Day 84
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The weighted mean FEV1 was derived by calculating the area under the curve, and then dividing the value by the relevant time interval. The weighted mean was calculated using the 6-hour serial FEV1 measurements at Day 84, which included pre-dose, and post-dose at 15 min, 30 min, 1 hour, 3 hours, and 6 hours. Baseline trough FEV1 is the mean of the two assessments made at -30 and -5 min pre-dose on Treatment Day 1. Change from Baseline was calculated as the Day 84 value minus the Baseline value. Analysis was performed using a repeated measures model with covariates of treatment, Baseline (mean of the two assessments made at -30and -5 min pre-dose on Treatment Day 1), smoking status, day, day by Baseline, and day by treatment interactions.
Time Frame: Baseline and Day 84
Population: ITT Population. Only those participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo QD + FSC 250/50 µg BID | UMEC 62.5 µg QD + FSC 250/50 µg BID | UMEC 125 µg QD + FSC 250/50 µg BID
Number analyzed (Participants) | 171 | 178 | 184
Liters | 0.052 (0.0137) | 0.196 (0.0135) | 0.217 (0.0133)

3. Secondary Outcome: Change From Baseline in the Mean Percentage of Rescue-free Days Over Weeks 1-12
Description: A rescue-free day is defined as a day on which no rescue medication was taken. Baseline calculations include a period of the later of 27 days before Visit 2 and the day after Visit 1, up to and including Day 1. The Weeks 1-12 calculations include a period from Study Day 2 up to the earlier of Study Day 85 and the day before Visit 7. Change from Baseline was calculated as the Weeks 1-12 value minus the Baseline value.
Time Frame: Baseline and Weeks 1- 12
Population: ITT Population. Only those participants available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Placebo QD + FSC 250/50 µg BID | UMEC 62.5 µg QD + FSC 250/50 µg BID | UMEC 125 µg QD + FSC 250/50 µg BID
Number analyzed (Participants) | 174 | 191 | 187
Percentage of days | 1.9 (27.38) | 8.4 (30.23) | 15.2 (28.25)

4. Secondary Outcome: Change From Baseline in the Mean Number of Puffs Per Day of Rescue Albuterol/Salbutamol Over Weeks 1-12
Description: The mean number of puffs per day of rescue albuterol/salbutamol at Baseline and on-treatment was recorded. The total puffs of rescue albuterol/salbutamol for each day was calculated as: (number of puffs + [2 * number of nebules]). Baseline calculations include a period of the later of 27 days before Visit 2 and the day after Visit 1, up to and including Day 1. The Weeks 1-12 calculations include a period from Study Day 2 up to the earlier of Study Day 85 and the day before Visit 7. Change from Baseline was calculated as the Weeks 1-12 value minus the Baseline value. Analysis was performed using an analysis of covariance (ANCOVA) model with covariates of treatment, Baseline (mean during the 4 weeks prior to Day 1), and smoking status.
Time Frame: Baseline and Weeks1- 12
Population: ITT Population. Only those participants available at the indicated time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: puffs
Arm/Group | Placebo QD + FSC 250/50 µg BID | UMEC 62.5 µg QD + FSC 250/50 µg BID | UMEC 125 µg QD + FSC 250/50 µg BID
Number analyzed (Participants) | 174 | 191 | 187
puffs | -0.2 (0.10) | -0.4 (0.10) | -0.7 (0.10)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) are defined as those events occurring while participants were on treatment or those events with an onset during the follow-up period (up to 13 weeks).
Description: SAEs and non-serious AEs are reported for members of the ITT Population, comprised of all participants randomized to treatment who received at least one dose of randomized study medication in the Treatment Period.
Arm/Group | Placebo QD + FSC 250/50 µg BID | UMEC 62.5 µg QD + FSC 250/50 µg BID | UMEC 125 µg QD + FSC 250/50 µg BID
Serious Adverse Events (participants affected / at risk) | 15/201 | 6/203 | 6/202
Other Adverse Events (participants affected / at risk) | 18/201 | 13/203 | 16/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD + FSC 250/50 µg BID (N=201) | UMEC 62.5 µg QD + FSC 250/50 µg BID (N=203) | UMEC 125 µg QD + FSC 250/50 µg BID (N=202)
Pneumonia (Infections and infestations) | 4 | 3 | 3
Infective exacerbation of chronic obstructive airways diseas (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD + FSC 250/50 µg BID (N=201) | UMEC 62.5 µg QD + FSC 250/50 µg BID (N=203) | UMEC 125 µg QD + FSC 250/50 µg BID (N=202)
Nasopharyngitis (Infections and infestations) | 9 | 6 | 10
Headache (Nervous system disorders) | 9 | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.